CLINICAL TRIAL: NCT02661477
Title: Clinical and Virological Efficacy of Pegylated Interferon Alpha in the Treatment of Rhinovirus Infection in Patients With Primary Hypogammaglobulinemia: Randomized Controlled Trial
Acronym: Hypogamma Int1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: T51/2015
Record Dates: First submitted 2016-01-13; First posted 2016-01-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Rhinovirus Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- pegylated interferon + placebo (Other): Patients with primary hypogammaglobulinemia and confirmed respiratory rhinovirus infection will receive subcutaneous pIFNα2a (pegylated interferon alfa 2, Pegasys, 180 ug s.c. injection once a week, two times ). Washout period is 8 weeks. When the same patient gets next rhinovirus infection, he/she will receive subcutaneous placebo (0,9% NaCl) injection once a week, two times.
  Interventions: Drug: pegylated interferon alfa 2; Other: Placebo
- placebo + pegylated interferon (Other): Patients with primary hypogammaglobulinemia and confirmed respiratory rhinovirus infection will receive will receivesubcutaneous placebo(0,9% NaCl) injection once a week, two times. Washout period is 8 weeks. When the same patient gets next rhinovirus infection, he/she will subcutaneous pIFNα2a (pegylated interferon alfa 2, Pegasys, 180 ug s.c. injection once a week, two times ).
  Interventions: Drug: pegylated interferon alfa 2; Other: Placebo

INTERVENTIONS:
Drug: pegylated interferon alfa 2
Other: Placebo — 0,9% natrium chlorine solution

SUMMARY:
The study will investigate the efficacy and safety of subcutaneous interferon alpha -2a to eradicate rhinovirus in patients with primary hypogammaglobulinemia. Patients with hypogammaglobulinemia have persistent rhinovirus infections. Rhinovirus may worsen pulmonary complications. Pegylated interferon alpha with ribavirin appear to effectively clear persistent rhinovirus infections in hypogammaglobulinemia patients.

Patients with primary hypogammaglobulinemia and confirmed respiratory rhinovirus infection will be randomly assigned in a double-blind fashion to receive either

* Group 1: subcutaneous pIFNα2a
* Group 2: subcutaneous placebo Subjects will have scheduled study visits at 1-week and at 2-month after entry to study. In addition, possible bacterial infections will be treated with antibiotics. Each patient will be followed with weekly nasal surveillance samples for 2 months and a symptom diary. Blood draws take place at study entry, 1-week and 2-month time-points.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years),
* primary hypogammaglobulinemia with regular immunoglobulin replacement therapy,
* rhinovirus positive from nasal swab,
* thrombocytes over 90 x109/L,
* Neutrophiles > 1,5 x109/L
* written informed consent.

Exclusion Criteria:

* Participation to another study,
* need for intensive care unit treatment,
* difficulties to understand national language, pregnancy and breastfeeding,
* any somatic, psychiatric or social disease or issue which in the opinion of the investigator makes participation in the trial not being in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Duration of respiratory symptoms | within 2 months
eradication of rhinovirus from nasal secretion (nasal secretion sample analyzed by rhinovirus PCR) | within 2 months (sample taken daily for 7 days, then weekly for 7 weeks)
time to next respiratory infection | within 2 months

SECONDARY OUTCOMES:
duration of respiratory symptoms | 2 months
  daily questionnaire for 8 weeks
rhinovirus genotype-specific persistence | 2 months
adverse events | 2 months
  symptom diary
blood counts | 2 months
  at time points 0, 1 wk and 2 months
alanine aminotransferase | 2 months
  at time points 0, 1 wk and 2 months
creatinine | 2 months
  at time points 0, 1 wk and 2 months
severity of respiratory functions | 2 months
  daily questionnaire for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Jartti, MD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku university hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No